CLINICAL TRIAL: NCT01945671
Title: The Influence of Obesity on Oocyte Functioning and Fertilization, Cumulus and Granulosa Functioning and Metabolic Factors.
Brief Title: The Influence of Obesity on Oocyte, Cumulus and Granulosa Functioning
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC 0070-13
Record Dates: First submitted 2013-09-15; First posted 2013-09-18 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-08

CONDITIONS: BMI; Lipid Profile

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. triglycerides, free fatty acid, cholesterol (HDl, LDL), insulin, glucose, lactate, IGF-1, Leptin E2, Progessterone, IL-1, Il-6 and TNF-2. α.blood free fluid from the leading follicle will be collected in a container for further evaluation of metabolic markers including triglycerides, free fatty acid, cholesterol (HDl, LDL), insulin, glucose, lactate, IGF-1, Leptin E2, Progessterone, IL-1, Il-6 and TNF-α , ROS.
  3. Cumulus cells 4. Oocytes diameter 5. GV oocytes, M1 and M2 that fail to fertilize 6. GDF-9, BMP-15, BMP-6, TNF-α, SMAD family will be analyzed by western blott as marker for oocytes quality.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Obese women have a higher prevalence of infertility than their lean counterparts. Obesity is a risk factor for anovulation , including in response to gonadotropin treatment .Further, even in women who are cycling regularly, obesity is associated with increased time-to-pregnancy and decreased chance of natural pregnancy.

During obesity or periods of overnutrition, lipid accumulates in nonadipose tissues, notably skeletal muscle, liver, heart, and pancreas due to cellular uptake of exogenous fatty acids, triglycerides, and cholesterol as well as de novo lipogenesis in response to elevated glucose. The accumulation of intracellular lipid leads to high levels of free fatty acids that are subject to oxidative damage and the formation of cytotoxic and highly reactive lipid peroxides, which ultimately are detrimental to intracellular organelles, particularly the endoplasmic reticulum (ER) and mitochondria. Exposure of the ER to high levels of free fatty acids and lipid peroxides causes structural alterations that perturb ER function and lead to accumulation of unfolded proteins and calcium release. Failure of the UPR to reestablish ER homeostasis can lead to apoptosis .When mitochondria are exposed to high levels of free fatty acids, these can become oxidized by mitochondrial reactive oxygen species, forming lipid peroxides that damage essential proteins and uncouple mitochondrial function. This results in mitochondrial damage, which can cause further accumulation of lipids that cannot be catabolized, disrupted cellular homeostasis, and ultimately apoptosis .

The cellular mechanisms by which obesity causes decreased conception rates are not known. Based on extensive evidence of obesity-induced lipotoxicity in other cells, it was hypothesized that obesity results in the activation of lipotoxicity pathways in the ovary. It was shown that lipid accumulation, ER stress, mitochondrial dysfunction, and apoptosis occur in ovarian cells and the oocyte in response to a high-fat diet.

The aim of our study was to evaluate the influence of high BMI on oocytes, granulose cells and metabolites in the follicular fluid.

DETAILED DESCRIPTION:
All women undergone IVF-ICSI cycles will be recruited in the study. They will be divided into 3 subgroups according to their BMI: 18.5-24.9 -normal; 25-29.9 - overweight ; ≥30 - obese.

i. A blood sample will be collected on the day of OPU and several markers will be checked- triglycerides, free fatty acid, cholesterol (HDl, LDL), insulin, glucose, lactate, IGF-1, Leptin E2, Progessterone, IL-1, Il-6 and TNF-α.

ii. After isolation of the oocytes from the follicular fluids - a blood free fluid from the leading follicle will be collected in a container for further evaluation of metabolic markers including triglycerides, free fatty acid, cholesterol (HDl, LDL), insulin, glucose, lactate, IGF-1, Leptin E2, Progessterone, IL-1, Il-6 and TNF-α , ROS.

iii. Cumulus cells will be collected after denudation of oocytes for ICSI and will be analyzed for apoptosis marker - Caspase 3 staining , Tunnel iv. Oocytes diameter - all denudated oocytes will be captured in the inverted microscope and the diameter will be measured.

v. GV oocytes, M1 and M2 that fail to fertilize will be analyzed for triglycerides, FFA and cholesterol concentration.

vi. GDF-9, BMP-15, BMP-6, TNF-α, SMAD family will be analyzed by western blott as marker for oocytes quality.

vii. Number of oocytes, mature (M2) oocytes, fertilization rate, cleavage rate, number embryos transferred, implantation rate, and pregnancy rate will be followed as well.

ELIGIBILITY:
Inclusion Criteria:

* All patients

Exclusion Criteria:

Ages: 20 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients undergo IVF treatments
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-01 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
pregnancy rate | 1 year

SECONDARY OUTCOMES:
lipid profile in different BMI | 1 year